CLINICAL TRIAL: NCT01698892
Title: Comparison of Respiratory Tolerance to I.V. Versus Sublingual Sedation During Bronchoscopy.
Brief Title: Comparison of Respiratory Tolerance to I.V. Versus Sublingual Sedation During Bronchoscopy. (TORSIV)
Acronym: TORSIV
Status: Terminated | Phase: Phase 4 | Type: Interventional
Why Stopped: End study
Sponsor: Nantes University Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: RC12_0208
Record Dates: First submitted 2012-10-01; First posted 2012-10-03 (Estimated); Last update posted 2023-11-18 (Actual); Status verified 2015-06

CONDITIONS: Sedation During Bronchoscopy
Keywords: I.V. sedation, midazolam, bronchoscopy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- I.V. sedation (Experimental): Patients who will undergo bronchoscopy will be followed during one day. They will be randomized in the I.V. sedation
  Interventions: Drug: I.V Sedation
- sublingual sedation (Active Comparator): Patients who will undergo bronchoscopy will be followed during one day. They will be randomized in the sublingual sedation group
  Interventions: Drug: sublingual sedation

INTERVENTIONS:
Drug: I.V Sedation — Patients who will undergo bronchoscopy will be followed during one day. They will be randomized in the I.V. sedation group
  Arms: I.V. sedation
Drug: sublingual sedation — Patients who will undergo bronchoscopy will be followed during one day. They will be randomized in the sublingual sedation group
  Arms: sublingual sedation

SUMMARY:
Bronchoscopy is a technique which currently allows the investigation of many respiratory diseases (infections, neoplasia, inflammation…) as well as endobronchial therapeutic procedures.

Good flexible bronchoscopy diagnostic practices suggest the use of anxiolytic premedication before endoscopy, but practices concerning the use of sedation further to the completion of the endoscopy are very heterogeneous.

We thus propose to compare, during a randomize, controlled trial, respiratory tolerance to I.V. versus sublingual sedation in two groups of patients indergoing bronchoscopy

ELIGIBILITY:
Inclusion Criteria:

* Men or women aged between 18 and 80, who will undergo bronchoscopy
* FEV1≥ 50% of theorical value
* Ambient air saturation at rest ≥ 94%
* No allergy to midazolam, to hydroxyzine, Lidocaine (used for local anesthesia) or one of their compound
* fasting for at least 6 hours
* No indication against bronchoscopy, nor to premedication
* Informed consent signed

Exclusion Criteria:

* Pregnant or lactating, women
* PAH patients
* patients undergoing bronchoscopy with bronchoalveolar lavage and / or trans-bronchial biopsy
* Patients with oral anticoagulants

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 85 (Actual)
Dates: Start 2012-10; Primary Completion 2014-12 (Actual); Study Completion 2014-12 (Actual)

PRIMARY OUTCOMES:
Intensity of dyspnea | 1 day
  Intensity of dyspnea assessed by the patient 1h after bronchoscopy in both groups measured by VAS (visual analogue scale) score (in millimeters on a 0 to 100 scale).

SECONDARY OUTCOMES:
VAS Individual scores | 1 day
  VAS Individual scores performed 1 hour after bronchoscopy (cough, nausea, pain, anxiety, overall tolerance)
Blood pressure | 1 day
  Blood pressure (mean blood pressure measurements made before, during and after the exam)
Desaturation frequency | 1 day
  Desaturation frequency during bronchoscopy, defined by the lowering of transcutaneous oxygen saturation below 90%
heart rate | 1 day
  Initial and maximum heart rate during bronchoscopy (continuous monitoring)
OAAS Score | 1 day
  OAAS Score after bronchoscopy
Bronchoscopy duration | 1 day
  Bronchoscopy duration (time difference between the input and output of the examination room, and between the start and end of bronchoscopy)
Comparison of midazolam total dose | 1 day
  Comparison of midazolam total dose administered in each group

CONTACTS AND LOCATIONS:
Locations (1):
- Cavailles, Nantes, France